CLINICAL TRIAL: NCT06241170
Title: Mesentery Guided Bowel Resection Margin Versus Traditional Margin in Reducing Early Endoscopic Recurrence Rate After Ileocolic Resection in Patients With Crohn 's Disease:a Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: Mesenteric Surgical Margin for Crohn's Disease Endoscopic Recurrence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Jinling Hospital, China (Other); Sir Run Run Shaw Hospital (Other); Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Jia Ke, Small Intestinal Surgery, Department of General Surgery, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZSLYEC-159
Record Dates: First submitted 2023-11-08; First posted 2024-02-05 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Endoscopic Recurrence Rate; After Ileocolic Crohn 's Disease Surgery
Keywords: endoscopic recurrence rate; ileocolic Crohn 's disease surgery; Mesentery Guided Resection

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mesentery-guided resection margin group (Experimental): Patients will undergo surgery using the mesentery-guided resection margin approach.
  Interventions: Procedure: mesentery-guided resection margin
- traditional resection margin group (Active Comparator): Patients will undergo surgery using the traditional resection margin approach.
  Interventions: Procedure: traditional resection margin

INTERVENTIONS:
Procedure: mesentery-guided resection margin — Mesentery-guided resection margin where the mesentery adjacent to the intestine completely transitions from abnormal to normal upon palpation and transillumination, compared to the proximal normal mesentery. Open, laparoscopic, hand-assisted, or robotic mobilization are all acceptable, but extracorporeal resection and anastomosis are required. After intestinal mobilization , the diseased intestinal segment is exteriorized from the abdominal cavity.
  Arms: mesentery-guided resection margin group
Procedure: traditional resection margin — 2 cm proximal to the site where gross lesions disappear. After transecting the bowel, re-examine the mucosal condition; if mucosal ulcers or obvious scars are present, extend the incision until reaching the site with normal mucosa. Definition of gross lesions: Evaluation from the outer intestinal wall: The site where the tough texture, thickening, or contracture at the mesenteric edge of the intestinal wall disappears; evaluation from the intestinal lumen: The site where mucosal ulcers, fissures, or obvious scars disappear. "Mucosa appearing seemingly abnormal" is considered normal.
  Arms: traditional resection margin group

SUMMARY:
Despite significant advancements in the treatment of Crohn's disease (CD), approximately 50% of patients undergo surgical intervention within ten years of diagnosis. Furthermore, more than 70% of these patients experience endoscopic recurrence within one year after surgery. This subset of patients often faces a poorer long-term prognosis and requires long-term intensified medical therapy. Therefore, reducing early postoperative endoscopic recurrence has remained a crucial focus in CD research.

From a surgical perspective, there have been limited breakthroughs in improving surgical techniques to reduce the postoperative endoscopic recurrence rate in CD. Recent research indicates that microscopic inflammation at the cut edge of the CD bowel segment is a significant risk factor for postoperative endoscopic recurrence. Mesenteric wrapping is a unique clinical pathological feature of CD. Our retrospective data suggest a clear linear correlation between the degree of mesenteric wrapping and microscopic inflammation in the corresponding bowel segment. Surgical margins determined by mesenteric guidance significantly reduce the postoperative endoscopic recurrence rate and clinical relapse rate compared to the traditional 2 cm margin. However, there is currently no prospective study comparing the efficacy of these two surgical approaches.To address this, investigators plan to conduct a multicenter randomized controlled trial. This trial will focus on patients with ileocolonic CD who have undergone primary anastomosis without residual disease. investigators aim to compare the postoperative endoscopic recurrence rates between mesenteric-guided margins and the traditional 2 cm margins. Our goal is to determine whether mesenteric-guided margins can reduce the postoperative endoscopic recurrence rate and to conduct relevant mechanistic research. Ultimately, this research may lead to the development of a novel surgical approach for CD based on the findings of this study.

DETAILED DESCRIPTION:
Current Status of the Study Current Status of the Study While treatment methods for Crohn's disease (CD) have made significant advancements, there is still a 50% requirement for surgical intervention within 10 years of diagnosis (1). The most common surgical procedures include ileocecal or terminal ileal resection. However, post-surgery, the risk of recurrence remains high, with 35% to 85% of patients experiencing endoscopic recurrence within one year (2, 4), and clinical recurrence occurring in 10% to 38% of patients within one year, leading to a need for reoperation in 30% of patients within five years (2, 3). Several studies have demonstrated that early endoscopic recurrence at six months post-surgery can effectively predict long-term treatment outcomes and guide subsequent medication choices (5).

Therefore, reducing early endoscopic anastomotic recurrence post-surgery has been a focus of CD research. The quality of surgical procedures significantly impacts this outcome. Previous research has identified risk factors for post-surgical recurrence, including smoking history, previous bowel resections, penetrating disease, extensive involvement, and concomitant perianal disease (6-8). However, these are non-modifiable patient-related factors. Within the scope of what physicians can control, proactive preventive treatment approaches adopted by gastroenterologists have been shown to reduce endoscopic recurrence rates to some extent. Nevertheless, the role and responsibilities of surgeons in this regard have not been clearly defined, and thus, there is a lack of standardized surgical strategies to reduce early endoscopic recurrence.（11） Intestinal mesentery abnormal proliferation and wrapping around the mesenteric margin is a characteristic pathological feature of Crohn's disease (CD). Recent studies have shown that mesenteric fat plays a crucial role in the development of CD (13, 14). The applicant's research team has also discovered the presence of bacteria displaced from the intestines within the mesentery, which can stimulate the proliferation of fat cells (15). Our preliminary retrospective data (pending submission) also suggests that if the mesenteric-guided margin, corresponding to the border of mesenteric abnormality, is used as the resection margin, even though an average of 10cm more intestine is removed, the postoperative endoscopic recurrence rate and clinical recurrence rate are significantly better than those of patients with the traditional limited 2cm margin (as described in the research foundation). However, there is currently no prospective randomized controlled study comparing these two margin strategies. Therefore, investigators plan to conduct a prospective multicenter randomized controlled study for patients with ileocolonic CD who undergo primary anastomosis without residual disease, comparing the postoperative endoscopic recurrence rates between mesenteric-guided margins and traditional 2cm margins, and conducting related mechanistic research to establish a high-level evidence for surgical margins that can reduce postoperative endoscopic recurrence in CD.

The significance of this research lies in addressing the issue of high endoscopic recurrence rates following surgery for Crohn's disease (CD), for which there is currently no established surgical solution. This study employs an innovative approach by using the mesenteric fat boundary as guidance for surgical resection margins, making it a novel contribution to both national and international research.

Building upon prior preliminary research, our research team aims to determine, through a prospective multicenter study, whether the use of mesentery-guided resection margins can reduce the endoscopic recurrence rate, while also exploring potential underlying mechanisms. The successful implementation of this project can provide high-level evidence for the correct selection of surgical margins in CD, fostering the development of personalized and precision surgical approaches in the treatment of CD in China, offering substantial clinical application and practical guidance.The ultimate goal of this study is to improve the long-term prognosis of CD patients and enhance their postoperative .

ELIGIBILITY:
Inclusion criteria:

1. Patients with a clear diagnosis of CD who meet the surgical indications and will undergo one-stage ileocecal resection,
2. Ileocecal CD with localized lesions involving the terminal ileum and cecum, with a total lesion length of <80 cm,
3. No residual lesions within 50 cm proximal to the ileocecal anastomosis,
4. Patients or their legal guardians who can understand and are willing to participate in this study, provide written informed consent, and have the ability to comply with the protocol.

Exclusion criteria:

1. Patients with a history of ileocecal resection,
2. Patients with primary lesions in other locations (e.g., proximal small bowel) that require surgical resection of inflamed intestinal segments other than the ileocecal region (excluding cases with affected other segments of the bowel),
3. Patients with a risk of short bowel syndrome,
4. Patients who require ileostomy formation,
5. Patients with severe anorectal lession,
6. Patients predicted to be unable to receive postoperative drug therapy,
7. Patients unable to return to the hospital for re-examination in a timely manner
8. Patients who have suffered from serious illnesses within the six months before surgery, such as myocardial infarction, active angina pectoris, congestive heart failure, or other diseases believed by the investigator to pose a risk to the patient's safety,
9. Patients with a history of malignant tumors, including melanoma (excluding localized skin cancer),
10. Patients clinically diagnosed with autoimmune diseases other than CD or with evidence of other autoimmune diseases.
11. Pregnant or lactating patients.
12. Patients who cannot be tracked at various study time points for the primary outcome measure.

Withdrawal criteria:

1. Subjects lost to follow-up or voluntarily requesting withdrawal.
2. The occurrence of anastomotic fistula after surgery that affects subsequent endoscopic evaluation.
3. Subjects considered unsuitable for further participation in the study by the investigator.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 172 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
The Modified Rutgeerts Score during colonoscopy | At 6 months after surgery.
  A Rutgeerts score > i2b is defined as endoscopic recurrence. Calculate the endoscopic recurrence rates in both groups and compare them using a chi-square test to determine if there is a significant difference between the two groups.

SECONDARY OUTCOMES:
To calculate the endoscopic recurrence rate for both groups within 1 year | At 1 year after surgery.
  Endoscopic Recurrence Rate = (Number of Patients with Endoscopic Recurrence / Total Number of Patients in the Group) * 100. Compare the recurrence rates between the two groups and determine if there is a significant difference, you can perform a chi-squared test.
Compare the postoperative margin pathology between the two surgical methods. | At 7 days after surgery
  In both the mesentery-guided margin and traditional limited resection specimens, within the range of 5-10 cm from the near margin (or up to the location of the diseased bowel segment), full-thickness pathological slides were taken every 1-2 cm (including the parts adjacent to the bowel mesentery) to assess if there is submucosal inflammation in the locations close to the macroscopic lesion and mesenteric abnormality.
Comparison of the length of bowel resection between the two surgical methods | At 7 days after surgery
  Calculate the average length of bowel resection in both groups and use a t-test to compare if there is a significant difference in resection length between the two groups.
Compare the clinical recurrence rates between the two groups | At 3 year after surgery.
  After the surgery, patients are required to undergo Crohn's Disease Activity Index (CDAI) scoring every 6 months. Patients with a CDAI score ≥150 are defined as experiencing clinical relapse. Clinical relapse rates for both groups are calculated (number of patients with clinical relapse in each group divided by the total number of patients in each group). A chi-squared test is then employed to compare if there are any differences in relapse rates between the two groups.
Calculate the rate of requiring a second surgery for both groups | At 3 years after surgery.
  Second surgery rate (number of individuals requiring a second surgery in each group divided by the total number in each group), and use the chi-squared test to compare whether there is a difference in the recurrence rates between the two groups.
Comparison of the intestinal function of paticipants between the two surgical methods | At 3 years after surgery.
  Evaluate postoperative bowel function using the GSRS scale, and require participants to complete the GSRS assessment every 6 months after surgery. Calculate the average GSRS scores in both groups and compare if there is a significant difference in GSRS scores between the two groups
Postoperative morbidity | A 30 days after surgery
  Morbidity according to the Clavien-Dindo classification，assessed 30 days after the two surgical techniques, included anastomotic leak、length of hospital stay，etc

CONTACTS AND LOCATIONS:
Overall Officials: Jia Ke, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Jia Ke, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Frolkis AD, Dykeman J, Negron ME, Debruyn J, Jette N, Fiest KM, Frolkis T, Barkema HW, Rioux KP, Panaccione R, Ghosh S, Wiebe S, Kaplan GG. Risk of surgery for inflammatory bowel diseases has decreased over time: a systematic review and meta-analysis of population-based studies. Gastroenterology. 2013 Nov;145(5):996-1006. doi: 10.1053/j.gastro.2013.07.041. Epub 2013 Jul 27. PMID 23896172
- [Background] Buisson A, Chevaux JB, Allen PB, Bommelaer G, Peyrin-Biroulet L. Review article: the natural history of postoperative Crohn's disease recurrence. Aliment Pharmacol Ther. 2012 Mar;35(6):625-33. doi: 10.1111/j.1365-2036.2012.05002.x. Epub 2012 Feb 7. PMID 22313322
- [Background] Frolkis AD, Lipton DS, Fiest KM, Negron ME, Dykeman J, deBruyn J, Jette N, Frolkis T, Rezaie A, Seow CH, Panaccione R, Ghosh S, Kaplan GG. Cumulative incidence of second intestinal resection in Crohn's disease: a systematic review and meta-analysis of population-based studies. Am J Gastroenterol. 2014 Nov;109(11):1739-48. doi: 10.1038/ajg.2014.297. Epub 2014 Oct 21. PMID 25331349
- [Background] Olaison G, Smedh K, Sjodahl R. Natural course of Crohn's disease after ileocolic resection: endoscopically visualised ileal ulcers preceding symptoms. Gut. 1992 Mar;33(3):331-5. doi: 10.1136/gut.33.3.331. PMID 1568651
- [Background] De Cruz P, Kamm MA, Hamilton AL, Ritchie KJ, Krejany EO, Gorelik A, Liew D, Prideaux L, Lawrance IC, Andrews JM, Bampton PA, Gibson PR, Sparrow M, Leong RW, Florin TH, Gearry RB, Radford-Smith G, Macrae FA, Debinski H, Selby W, Kronborg I, Johnston MJ, Woods R, Elliott PR, Bell SJ, Brown SJ, Connell WR, Desmond PV. Crohn's disease management after intestinal resection: a randomised trial. Lancet. 2015 Apr 11;385(9976):1406-17. doi: 10.1016/S0140-6736(14)61908-5. Epub 2014 Dec 24. PMID 25542620
- [Background] Auzolle C, Nancey S, Tran-Minh ML, Buisson A, Pariente B, Stefanescu C, Fumery M, Marteau P, Treton X, Hammoudi N; REMIND Study Group Investigators; Jouven X, Seksik P, Allez M. Male gender, active smoking and previous intestinal resection are risk factors for post-operative endoscopic recurrence in Crohn's disease: results from a prospective cohort study. Aliment Pharmacol Ther. 2018 Nov;48(9):924-932. doi: 10.1111/apt.14944. Epub 2018 Aug 20. PMID 30126030
- [Background] Magro F, Gionchetti P, Eliakim R, Ardizzone S, Armuzzi A, Barreiro-de Acosta M, Burisch J, Gecse KB, Hart AL, Hindryckx P, Langner C, Limdi JK, Pellino G, Zagorowicz E, Raine T, Harbord M, Rieder F; European Crohn's and Colitis Organisation [ECCO]. Third European Evidence-based Consensus on Diagnosis and Management of Ulcerative Colitis. Part 1: Definitions, Diagnosis, Extra-intestinal Manifestations, Pregnancy, Cancer Surveillance, Surgery, and Ileo-anal Pouch Disorders. J Crohns Colitis. 2017 Jun 1;11(6):649-670. doi: 10.1093/ecco-jcc/jjx008. No abstract available. PMID 28158501
- [Background] Fumery M, Dulai PS, Meirick P, Farrell AM, Ramamoorthy S, Sandborn WJ, Singh S. Systematic review with meta-analysis: recurrence of Crohn's disease after total colectomy with permanent ileostomy. Aliment Pharmacol Ther. 2017 Feb;45(3):381-390. doi: 10.1111/apt.13886. Epub 2016 Dec 8. PMID 27928830
- [Background] Fazio VW, Marchetti F, Church M, Goldblum JR, Lavery C, Hull TL, Milsom JW, Strong SA, Oakley JR, Secic M. Effect of resection margins on the recurrence of Crohn's disease in the small bowel. A randomized controlled trial. Ann Surg. 1996 Oct;224(4):563-71; discussion 571-3. doi: 10.1097/00000658-199610000-00014. PMID 8857860
- [Background] Riault C, Diouf M, Chatelain D, Yzet C, Turpin J, Brazier F, Dupas JL, Sabbagh C, Nguyen-Khac E, Fumery M. Positive histologic margins is a risk factor of recurrence after ileocaecal resection in Crohn's disease. Clin Res Hepatol Gastroenterol. 2021 Sep;45(5):101569. doi: 10.1016/j.clinre.2020.10.013. Epub 2020 Nov 14. PMID 33199239
- [Background] Tandon P, Malhi G, Abdali D, Pogue E, Marshall JK, de Buck van Overstraeten A, Riddell R, Narula N. Active Margins, Plexitis, and Granulomas Increase Postoperative Crohn's Recurrence: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2021 Mar;19(3):451-462. doi: 10.1016/j.cgh.2020.08.014. Epub 2020 Aug 12. PMID 32801016
- [Background] de Buck van Overstraeten A, Eshuis EJ, Vermeire S, Van Assche G, Ferrante M, D'Haens GR, Ponsioen CY, Belmans A, Buskens CJ, Wolthuis AM, Bemelman WA, D'Hoore A. Short- and medium-term outcomes following primary ileocaecal resection for Crohn's disease in two specialist centres. Br J Surg. 2017 Nov;104(12):1713-1722. doi: 10.1002/bjs.10595. Epub 2017 Jul 26. PMID 28745410
- [Background] Holt DQ, Moore GT, Strauss BJ, Hamilton AL, De Cruz P, Kamm MA. Visceral adiposity predicts post-operative Crohn's disease recurrence. Aliment Pharmacol Ther. 2017 May;45(9):1255-1264. doi: 10.1111/apt.14018. Epub 2017 Feb 28. PMID 28244124
- [Background] Li Y, Ge Y, Gong J, Zhu W, Cao L, Guo Z, Gu L, Li J. Mesenteric Lymphatic Vessel Density Is Associated with Disease Behavior and Postoperative Recurrence in Crohn's Disease. J Gastrointest Surg. 2018 Dec;22(12):2125-2132. doi: 10.1007/s11605-018-3884-9. Epub 2018 Jul 24. PMID 30043133
- [Background] He Z, Wu J, Gong J, Ke J, Ding T, Zhao W, Cheng WM, Luo Z, He Q, Zeng W, Yu J, Jiao N, Liu Y, Zheng B, Dai L, Zhi M, Wu X, Jobin C, Lan P. Microbiota in mesenteric adipose tissue from Crohn's disease promote colitis in mice. Microbiome. 2021 Nov 23;9(1):228. doi: 10.1186/s40168-021-01178-8. PMID 34814945